CLINICAL TRIAL: NCT01072682
Title: A Multi-Center Pilot Study to Assess the Safety and Efficacy of A Selective Cytopheretic Device (SCD) Treatments In Patients With Acute Renal Failure (ARF)
Brief Title: Safety Study of a Selective Cytopheretic Device (SCD) in Patients With Acute Renal Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SeaStar Medical (Industry)
Collaborators: Baim Institute for Clinical Research (Other); Medtox (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARF002
Record Dates: First submitted 2010-02-17; First posted 2010-02-22 (Estimated); Results first posted 2022-03-09 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Acute Renal Failure
Keywords: Acute Renal Failure; Acute tubular necrosis; Continuous Renal Replacement Therapy; Selective cytopheretic device
MeSH Terms: conditions — Acute Kidney Injury; Kidney Cortex Necrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SCD (Experimental): Selective Cytopheretic Device
  Interventions: Device: Selective cytopheretic device (SCD)

INTERVENTIONS:
Device: Selective cytopheretic device (SCD) — The selective cytopheretic device (SCD) is comprised of tubing, connectors and a hemofilter cartridge. The device is connected in series to a commercially available Continuous Renal Replacement Therapy (CRRT) device. Blood from the CRRT circuit is diverted after the CRRT hemofilter through to the extra capillary space (ECS) of the SCD. Blood circulates through this space and is returned to the patient via the venous return line of the CRRT circuit. Regional citrate anticoagulation is used for the entire CRRT and SCD blood circuits.

SUMMARY:
The purpose of this protocol is to evaluate the safety of a selective cytopheretic device (SCD) in patients that are on continuous renal replacement therapy (CRRT) for acute renal failure (ARF).

DETAILED DESCRIPTION:
Acute renal failure is a condition where the kidneys are not capable of producing adequate urine. Therefore, another way to remove waste from the body is needed to hopefully allow time for the kidneys to heal. One method of removing waste from the body is called Continuous Renal Replacement Therapy (CRRT) or variations of that therapy. This study will evaluate the safety of the device while it is connected to the CRRT tubing for up to 7 days. Patients will be followed up until day 60 following the treatment.

ELIGIBILITY:
Inclusion Criteria:

1. A patient, or legal representative, has signed a written informed consent form.
2. Must be receiving medical care in an intensive care unit (e.g., ICU, MICU, SICU, CTICU, Trauma, Mixed, other).
3. Age 18 to 80 years.
4. Females of child bearing potential who are not pregnant (confirmed by a negative serum pregnancy test) and not lactating if recently post-partum.
5. Must be receiving and tolerating CRRT therapy for a minimum of 4 hours, but not longer than 24 hours.
6. Expected to remain in the ICU for at least 96 hours after evaluation for enrollment.
7. A clinical diagnosis of ATN due to hemodynamic or toxic etiologies. ATN is defined as acute renal failure occurring in a setting of acute ischemic or nephrotoxic injury with oliguria (average <20 mL/hr) for >6-12 hours or: an increase in serum creatinine ≥2 mg/dL (≥1.5 mg/dL in females) over a period of ≤4 days. (Note: Prerenal, hepatorenal, vascular, interstitial, glomerular, and obstructive etiologies are excluded on clinical or other diagnostic grounds.)
8. At least one non-renal organ failure (modified SOFA organ system score >2), as defined in Appendix A or presence (proven or suspected) of sepsis as defined in Appendix B.
9. All patients must be able to tolerate regional citrate anticoagulation.

Exclusion Criteria:

1. Contraindications to regional citrate anticoagulation.
2. Irreversible brain damage based on available historical and clinical information.
3. Presence of a renal transplant at any time.
4. Non-candidacy for acute renal replacement therapy.
5. Non-renal organ transplantation within six months of screening date.
6. Presence of preexisting chronic renal failure prior to this episode of ARF. Preexisting chronic renal failure is defined as baseline serum creatinine >2.5 mg/dL (men), or >2.0 mg/dL (women).
7. ARF occurring in the setting of burns, obstructive uropathy, allergic interstitial nephritis, acute or rapidly progressive glomerulonephritis, vasculitis, hemolytic-uremic syndrome, thrombotic thrombocytopenic purpura (TTP), malignant hypertension, scleroderma renal crisis, atheroembolism, functional or surgical nephrectomy, hepatorenal syndrome, cyclosporine or tacrolimus nephrotoxicity.
8. Metastatic malignancy which is actively being treated or may be treated by chemotherapy or radiation during the subsequent three month period after study therapy
9. Chronic immunosuppression (e.g., AIDS, chronic glucocorticoid therapy >20 mg/day prednisone equivalent on a chronic basis, or chemotherapy). The acute use of glucocorticoids is permissible
10. Severe liver failure as documented by a Child-Pugh Liver Failure Score >12.
11. Do Not Resuscitate (DNR) status.
12. Comfort measures only.
13. Patient is moribund or for whom full supportive care is not indicated.
14. Patient not expected to survive 28 days because of an irreversible medical condition.
15. Any medical condition that the Investigator thinks may interfere with the study objectives.
16. Physician refusal.
17. Patient pregnant.
18. Patient is a prisoner.
19. Pre-morbid weight >128.5 kg.
20. More than one hemodialysis treatment or longer than 24 hours since starting CRRT.
21. Platelet count <30,000/mm3.
22. Concurrent enrollment in another interventional clinical trial. Patients enrolled in clinical trials where only measurements and or samples are taken (NO TEST DEVICE OR DRUG USED) are allowed to participate.
23. Use of any other Investigational drug or device within the previous 30 days.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2010-02; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - University of Alabama Birmingham, Birmingham, Alabama
  - University of California San Diego, San Diego, California
  - Denver Nephrology, Denver, Colorado
  - George Washington University, Washington D.C., District of Columbia
  - Mayo Clinic, Rochester, Minnesota
  - Memorial Hospital, Chattanooga, Tennessee
  - University of Texas, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- SCD Experimental Treatment Arm: Selective Cytopheretic Device
  Selective cytopheretic device (SCD): The selective cytopheretic device (SCD) is comprised of tubing, connectors and a hemofilter cartridge. The device is connected in series to a commercially available Continuous Renal Replacement Therapy (CRRT) device. Blood from the CRRT circuit is diverted after the CRRT hemofilter through to the extra capillary space (ECS) of the SCD. Blood circulates through this space and is returned to the patient via the venous return line of the CRRT circuit. Regional citrate anticoagulation is used for the entire CRRT and SCD blood circuits.
Period: Overall Study
Arm/Group | SCD Experimental Treatment Arm
Started | 35
Completed | 35
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | SCD Experimental Treatment Arm
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.3 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 25
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 35

OUTCOME MEASURES:

1. Primary Outcome: 60 Day Mortality
Time Frame: Day 60 following treatment end
Measure: Count of Participants; unit: Participants
Arm/Group | SCD Experimental Treatment Arm
Number analyzed (Participants) | 35
Participants | 11

2. Primary Outcome: 60 Day Renal Recovery
Description: The criteria used to measure Renal Recovery requires the patient to be dependent free of CRRT and/or chronic dialysis.
Time Frame: Day 60 following treatment end
Population: Renal Recovery in surviving subjects at Day 60
Measure: Count of Participants; unit: Participants
Arm/Group | SCD Experimental Treatment Arm
Number analyzed (Participants) | 24
Participants | 24

ADVERSE EVENTS:
Arm/Group | SCD Experimental Treatment Arm
All-Cause Mortality (participants affected / at risk) | 11/35
Serious Adverse Events (participants affected / at risk) | 23/35
Other Adverse Events (participants affected / at risk) | 33/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SCD Experimental Treatment Arm (N=35)
Right Iliac Artery Injury (Vascular disorders) | 1 (1)
Complicated Abdominal Wound (Infections and infestations) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Septic Shock (Infections and infestations) | 1 (1)
Cardiogenic Shock (Cardiac disorders) | 1 (1)
Sepsis (Infections and infestations) | 3 (3)
Pneumonia (Infections and infestations) | 2 (2)
Hypocalcemia (Blood and lymphatic system disorders) | 1 (1)
Ventricular Fibrillation (Cardiac disorders) | 1 (1)
DIC (Blood and lymphatic system disorders) | 2 (2)
Multi-System Organ Failure (General disorders) | 3 (3)
Pulmonary Thromboembolism (Blood and lymphatic system disorders) | 1 (1)
GI Bleed (Gastrointestinal disorders) | 1 (1)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Chest Tube Bleed (Surgical and medical procedures) | 1 (1)
Empyema (Infections and infestations) | 1 (1) — Right Lung
Nutritional Deficiency (Metabolism and nutrition disorders) | 1 (1)
Multifactorial Anemia (Blood and lymphatic system disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Due to ventilator
Multiple Spontaneous Pneumothoraces (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Altered Mental Status (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SCD Experimental Treatment Arm (N=35)
Thrombocytopenia (Blood and lymphatic system disorders) | 9 (10)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2)
Hypotension (Cardiac disorders) | 7 (7)
Anemia (Blood and lymphatic system disorders) | 7 (7)
Leukocytosis (Metabolism and nutrition disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 4 (4)
Metabolic Alkalosis (Metabolism and nutrition disorders) | 2 (2)
Respiratory Alkalosis (Metabolism and nutrition disorders) | 3 (3)
Non-occlusive Thrombus (Blood and lymphatic system disorders) | 2 (2)
Candidiasis (Infections and infestations) | 4 (4)
Hypomagnesemia (Metabolism and nutrition disorders) | 4 (4)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Ventricular Tachycardia (Cardiac disorders) | 3 (3)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 5 (5)
Bradycardia (Cardiac disorders) | 2 (2)
Hypoglycemia (Endocrine disorders) | 2 (2)
Atrial Fibrillation (Cardiac disorders) | 4 (4)
Hematoma (General disorders) | 2 (2)
Rectal Bleed (Gastrointestinal disorders) | 4 (4)
Sepsis (Infections and infestations) | 3 (3)
Generalized Pain (General disorders) | 4 (4)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2)
Agitation (General disorders) | 4 (4)
Deep Vein Thrombosis (DVT) (Blood and lymphatic system disorders) | 3 (3)
Sinus Tachycardia (Cardiac disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Hypervolemia (General disorders) | 4 (4)
Pneumonia (Infections and infestations) | 2 (2)
Anxiety (Psychiatric disorders) | 2 (2)
Encephalopathy (General disorders) | 2 (2)
Ileus (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No